CLINICAL TRIAL: NCT01948037
Title: Hydrotherapy for the Treatment of Symptomatic Lower Extremity Arterial Disease in Diabetes Type 2 Patients:A Randomized Controlled Trial
Brief Title: Effectiveness Study of Hydrotherapy Against Pain and Other Symptoms in Diabetes-induced LEAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NanjingJH
Record Dates: First submitted 2013-09-13; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes; Lower Extremity Arterial Disease
Keywords: hydrotherapy; randomized controlled trial; lower extremity arterial disease; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Hydrotherapy; Hot Springs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrotherapy (Active Comparator)
  Interventions: Other: hydrotherapy
- hot spring (Other): 30-minutes/per day;4weeks
  Interventions: Other: hydrotherapy

INTERVENTIONS:
Other: hydrotherapy — 30-minutes/per day,for 4weeks
Other: hydrotherapy — 30-minutes/per day;4weeks
  Other Names: hot spring

SUMMARY:
The purpose of the study is to investigate whether the hydrotherapy are effective in against pain and other symptoms in diabetes-induced LEAD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes mellitus
* diagnosis of lower extremity arterial disease

Exclusion Criteria:

* Severe heart disease
* can't hydrotherapy

Ages: 48 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from the intensity of numbness and cold feeling at 4 weeks. Change from the improvement of the pain index at 4 weeks. | 4 weeks

SECONDARY OUTCOMES:
Change from ankle-brachial index at 4 weeks | 4 weeks

OTHER OUTCOMES:
Change from flow velocity values at 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Y bin, Study Chair — Jinling Hospital, China
Locations (1):
- Nanjing Jinling Hospital, Nanjing, Jiangsu, China